CLINICAL TRIAL: NCT01478009
Title: A Placebo-Controlled Trial of Korean Red Ginseng Extract to Prevent Acute Respiratory Illness in Healthy Subjects
Brief Title: Efficacy of an Extract of Concentrated Korean Red Ginseng for Preventing Upper Respiratory Tract Infections
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IJRG-INFL-KRG
Record Dates: First submitted 2011-11-16; First posted 2011-11-23 (Estimated); Results first posted 2012-12-25 (Estimated); Last update posted 2012-12-25 (Estimated); Status verified 2012-11

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Asian ginseng

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- KRG Extract (Experimental)
  Interventions: Dietary Supplement: Korean red ginseng
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Korean red ginseng — Korean red ginseng(3.0g/day) for 12 weeks
  Arms: KRG Extract
Dietary Supplement: Placebo — Placebo (3.0g/day) for 12 weeks
  Arms: Placebo

SUMMARY:
Upper respiratory tract infections are a major source of morbidity throughout the world. Extracts of Korean red ginseng have been found to have the potential to modulate both natural and acquired immune responses. The investigators sought to examine the efficacy of an extract of Korean red ginseng in preventing colds. Therefore, the efficacy and safety of Korean red ginseng will be investigated in healthy subjects during the influenza season.

DETAILED DESCRIPTION:
The extract of Korean red ginseng has been found efficacious in the prevention of respiratory infections in healthy adults. The investigators will be conducted a randomized, double-blind, placebo-controlled study at the onset of the influenza season. A total of 100 subjects 30-70 years of age with a history of at least 2 colds in the previous year will be recruited from the general population in jeollabuk-do, South Korea. The subjects will be instructed to take 9 capsules per day of either the Korean red ginseng extract or a placebo for a period of 12weeks. The primary outcome measure will be the number of Jackson-verified colds. Secondary outcome measures will be included symptom severity, total number of days of symptoms and duration of all colds. Cold symptoms will be scored by subjects.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 30-70 years old
* have contracted at least 2 colds in the past year

Exclusion Criteria:

* if they had been vaccinated against influenza in the previous 6 months.
* Subjects with medical conditions such as multiple sclerosis, tuberculosis, diabetes, cancer, lupus, HIV/AIDS, cardiovascular disease, hypertension, neurologic or psychiatric disease, and renal, pulmonary and hepatic abnormalities
* Subjects taking medications such as immunosuppressive drugs, corticosteroids, warfarin, phenalzine, pentobarbital, haloperidol or cyclosporine
* Abnormal liver or kidney function tests (ALT or AST>2 times the upper limit of normal; elevated creatinine, males>125uM/L, females>110uM/L)
* pregnant or lactating women and heavy smokers.
* being judged by the responsible physician of the local study center as unfit to participate in the study

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Seop Lee, MD, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Clinical Trial Center for Functional Foods; Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea

REFERENCES:
- [Derived] Lee CS, Lee JH, Oh M, Choi KM, Jeong MR, Park JD, Kwon DY, Ha KC, Park EO, Lee N, Kim SY, Choi EK, Kim MG, Chae SW. Preventive effect of Korean red ginseng for acute respiratory illness: a randomized and double-blind clinical trial. J Korean Med Sci. 2012 Dec;27(12):1472-8. doi: 10.3346/jkms.2012.27.12.1472. Epub 2012 Dec 7. PMID 23255845
- [Derived] Ha KC, Kim MG, Oh MR, Choi EK, Back HI, Kim SY, Park EO, Kwon DY, Yang HJ, Kim MJ, Kang HJ, Lee JH, Choi KM, Chae SW, Lee CS. A placebo-controlled trial of Korean red ginseng extract for preventing influenza-like illness in healthy adults. BMC Complement Altern Med. 2012 Feb 8;12:10. doi: 10.1186/1472-6882-12-10. PMID 22314101

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through local advertising and doctor referrals from hospital outpatients and general practice clinics.
Pre-assignment Details: The criteria were an age from 30 to 70 years, have contracted at least 2 colds in the past year. Subjects were excluded if they had been vaccinated against influenza in the previous 6 months.
Groups:
- KRG(Korean Red Ginseng) Extract: KRG Extract(3times/day, 9capsules/day, 3g/day) for 12weeks
  KRG Extract : KRG Extract was extracted at high temperatures (above 95℃)
- Placebo: Placebo(3times/day, 9capsules/day, 3g/day) for 12weeks
  Placebo : Amount and calorie of placebo are same with KRG Extract.
Period: Overall Study
Arm/Group | KRG(Korean Red Ginseng) Extract | Placebo
Started | 50 | 50
Completed | 49 | 49
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KRG Extract | Placebo | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 45.5 (8.1) | 46.3 (9.8) | 45.9 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 34 | 62
  Male | 22 | 16 | 38
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Frequency of ILI(Influenza Like Illness)
Description: Subjects received the open-ended questions about frequency of ILI onset during study period. The frequency of ILI onset was checked weekly via telephone.
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Number; unit: participants
Groups:
- KRG Extract: Oral intake Korean red ginseng(3.0g/day) for 12weeks.
- Placebo: Oral intake placebo(3.0g/day) for 12weeks
Arm/Group | KRG Extract | Placebo
Number analyzed (Participants) | 49 | 49
participants | 12 | 22

2. Secondary Outcome: Symptom Severity of All Colds
Description: Subjects received the open-ended questions about symptom severity of all colds onset during study period. The symptom severity of all colds onset was checked weekly via telephone.
  Symptom severity of all colds (score 0-27) was measured during study period. The original index consists of 9 Questions(Fever, Rhinorrhea, Nasal congestion, Sore throat, Cough, Sputum, Dyspnea, Headache, Myalgia).
  Individual question response is assigned a score of between 0 (none) to 3 (severe) and summed to form a total score(summed) ranging from 0 (best) to 27 (worst).
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | KRG Extract | Placebo
Number analyzed (Participants) | 49 | 49
Scores on a scale | 9.5 (4.5) | 17.6 (23.1)

3. Secondary Outcome: Total Number of Days of Symptoms and Duration of All Colds
Description: Extract of Korean red ginseng intake did not significantly reduced total number of days of symptoms and duration of all colds
Time Frame: up to 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Serious and/or other [non-serious] adverse events were not collected/assessed
Arm/Group | KRG Extract | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No